CLINICAL TRIAL: NCT06921928
Title: A Phase I/II Open-label Dose Escalation and Dose Expansion Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of AZD4360 in Adult Participants With Advanced Solid Tumours
Brief Title: Study for AZD4360 in Participants With Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8930C00001; 2024-518281-27-00 (Other: EU CT Number)
Record Dates: First submitted 2025-03-25; First posted 2025-04-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Gastric Cancer; Gastroesophageal Junction Cancer; Biliary Tract Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: Gastric Cancer; Gastroesophageal Junction Cancer; Biliary Tract Cancer; Pancreatic Ductal Adenocarcinoma; Advanced Solid Tumours; AZD4360; Claudin 18.2
MeSH Terms: conditions — Stomach Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AZD4360 Monotherapy (Experimental): AZD4360 Monotherapy
  Interventions: Drug: AZD4360

INTERVENTIONS:
Drug: AZD4360 — Antibody-Drug Conjugate targeting Claudin 18.2 (CLDN18.2)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, PK, immunogenicity, pharmacodynamics, and preliminary efficacy of AZD4360 in adult participants with locally advanced or metastatic solid tumours selected for expression of CLDN18.2.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 at the time of signing the ICF.
2. Eastern cooperative oncology group performance status of 0-1 with no deterioration over the previous 2 weeks prior to baseline or day of first dosing.
3. Minimum life expectancy of 12 weeks in the opinion of the Investigator.

4 Adequate organ and marrow function, as defined by protocol.

5. Contraceptive use by men or women should be consistent with local regulations, as defined by protocol.

6. Histologically confirmed advanced or metastatic Pancreatic ductal adenocarcinoma (PDAC), Gastric or Gastroesophageal junction cancer (G/GEJC), and Biliary tract cancer (BTC) with documented positive CLDN18.2 expression.

7. Participants must have received at least one prior line of systemic therapy in the advanced/metastatic disease.

8. At least one measurable lesion according to RECIST v1.1.

Exclusion Criteria:

1. Human Epidermal Growth Factor Receptor 2 (HER2) positive (3+ by IHC or 2+ by IHC and positive by in situ hybridisation) or indeterminate G/GEJC participants.
2. Unstable or active peptic ulcer disease or digestive tract bleeding including but not limited to clinically significant bleeding in the setting of prior CLDN18.2 directed therapy.
3. Participants with clinically significant ascites that require drainage.
4. Central nervous system (CNS) metastases or CNS pathology, as defined by protocol.
5. With spinal cord compression or with high risk of paralysis.
6. History of non-infectious interstitial lung disease/pneumonitis.
7. Participant has cardiac abnormalities, as defined by protocol.
8. History of another primary malignancy within 2 years prior to screening.
9. Known serologic status reflecting active hepatitis B or hepatitis C.
10. Known HIV infection that is not well controlled.
11. Active tuberculosis infection.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of participants with Dose-Limiting Toxicity (in dose escalation cohort), Adverse events (AEs) , Serious Adverse Events (SAEs) and AEs leading to discontinuation of AZD4360 | Through study completion, up to approximately 2 years
  To investigate the safety and tolerability, and to determine the Maximum Tolerated Dose (MTD) and/or a Recommended Phase II Dose (R2PD) of AZD4360 in previously treated participants with advanced solid tumours, through the assessment of Dose Limiting Toxicities, Adverse Events and Severe Adverse Events.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Through study completion, up to approximately 2 years
  The percentage of participants with a confirmed Complete Response (CR) or Partial Response (PR).
  Radiological response evaluated according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1.
Duration of Response (DoR) | Through study completion, up to approximately 2 years
  The time from the date of first documented ORR until date of first documented Progression of Disease (PD) or death.
  Radiological response evaluated according to RECIST v1.1.
Disease Control Rate (DCR) | Through study completion, up to approximately 2 years
  The percentage of participants who have a best objective response of confirmed CR or PR or who have Stable Disease for at least 11 weeks after start of treatment to allow for an early assessment within the assessment window.
  Radiological response evaluated according to RECIST v1.1.
Progression Free Survival (PFS) | Through study completion, up to approximately 2 years
  The time from the start of treatment until the date of objective PD or death.
  Radiological response evaluated according to RECIST v1.1.
Overall Survival (OS) | Through study completion, up to approximately 2 years
  The time from the start of treatment until death due to any cause.
Plasma pharmacokinetics (PK) parameters of AZD4360: Plasma concentration | Through study completion, up to approximately 2 years
  Plasma concentration of AZD4360, total antibody and other analytes.
Plamsa PK parameters of AZD4360, total antibody and other analytes: Area Under Curve (AUC) | Through study completion, up to approximately 2 years
  Area under the plasma concentration versus time curve for AZD4360, total antibody and other analytes.
Plasma PK parameters of AZD4360, total antibody and other analytes: Maximum plasma concentration (Cmax) | Through study completion, up to approximately 2 years
  Maximum observed plasma concentration of AZD4360, total antibody and other analytes.
Plasma PK parameters of AZD4360, total antibody and other analytes: Time to maximum plasma concentration (tmax) | Through study completion, up to approximately 2 years
  The time it takes for AZD4360, total antibody and other analytes to reach the maximum plasma concentration after administration of the study drug.
Plasma PK parameters of AZD4360, total antibody and other analytes: Clearance | Through study completion, up to approximately 2 years
  A pharmacokinetic measurement of the volume of plasma from which AZD4360, total antibody and other analytes are completely removed per unit time.
Plasma PK parameters of AZD4360, total antibody and other analytes: Half-life | Through study completion, up to approximately 2 years
  The time required for the quantity of AZD4360, total antibody and other analytes to reduce to half of their initial values.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (3):
  - Research Site, Santa Monica, California
  - Research Site, Providence, Rhode Island
  - Research Site, Houston, Texas
- China (4):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Shanghai
  - Research Site, Wuhan
- Germany (3):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Frankfurt
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Kashiwa
  - Research Site, Kōtoku
- United Kingdom (2):
  - Research Site, Glasgow
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/